CLINICAL TRIAL: NCT00000137
Title: Collaborative Corneal Transplantation Studies (CCTS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-36
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Corneal Transplantation; Graft Rejection

INTERVENTIONS:
Procedure: Histocompatibility Matching

SUMMARY:
To determine whether histocompatibility matching of corneal transplant donors and recipients can reduce the incidence of graft rejection in high-risk patients.

DETAILED DESCRIPTION:
Approximately 20 percent of corneal transplant patients, about 6,000 per year, face donor tissue rejection at rates of up to 60 percent because of corneal vascularization or prior graft rejection. Histocompatibility antigen matching and/or crossmatching may have offered these patients an improved chance for successful outcome.

The Collaborative Corneal Transplantation Studies Group conducted two controlled, double-masked studies addressing distinct scientific questions about donor-recipient histocompatibility matching. The Crossmatch Study was a randomized study assessing the effectiveness of crossmatching in preventing graft rejection among high-risk patients with lymphocytotoxic antibodies. The Antigen Matching Study was a prospective, double-masked, observational study of the effectiveness of HLA-A, -B, and -DR donor-recipient matching in high-risk patients who had no lymphocytotoxic antibodies.

Six clinical centers recruited high-risk patients and collaborated with their local eye banking and organ procurement agencies in procuring donor corneal tissue. For each of the two studies, a total of 400 patients were sought. Blood samples from each enrolled patient were sent to the local CCTS tissue typing laboratory for HLA typing, and serum samples were sent to the Central Laboratory to be screened for preformed lymphocytotoxic antibodies. Depending on the results of the testing, patients were entered into the Crossmatch Study or the Antigen Matching Study.

As corneal donors became available, donor blood samples were HLA typed at the local laboratories and crossmatched against all CCTS patients who awaited transplantation. Results of the testing were entered in a national, 24-hour computerized allocation system operated by the United Network for Organ Sharing (UNOS). Patients in the Crossmatch Study received a cornea from either a positively crossmatched donor or a negatively crossmatched donor. Patients in the Antigen Matching Study received a cornea with 0 to 6 matched antigens.

Transplant patients were followed intensively during the first months after surgery. The number of clinic visits was tapered to 2 during the third and final year of followup, resulting in a total of 17 postoperative visits. Irreversible failure of the corneal allograft due to all causes was the primary outcome variable in both studies. Allograft reaction episodes, irreversible failure due to rejection, and visual acuity were secondary outcome variables.

ELIGIBILITY:
Males and females age 10 years or older with two to four quadrants of corneal stroma vascularization or a history of allograft rejection in the eye considered for surgery were eligible for both studies in the CCTS.

Patients must have been willing to participate in 3 years of followup. No one was eligible for the CCTS who had a condition that would greatly increase the risk of nonrejection graft failure, such as xerophthalmia or severe exposure keratopathy. Also excluded were patients with systemic diseases or with medication usage that might alter their immune response.

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-05; Study Completion 1989-09 (Actual)

REFERENCES:
- [Background] Stark WJ, Stulting RD, Thoft R. HLA matching and corneal transplantation. N Engl J Med. 1987 Dec 3;317(23):1476-7. doi: 10.1056/NEJM198712033172311. No abstract available. PMID 3317044
- [Background] Klein PK; Stark WJ; Maguire MG; Stulting RD; Collaborative Corneal Transplantation Research Group; Donor-recipient crossmatching and typing to avoid corneal allograft rejection, in Cavanaugh HD (ed)., The Cornea: The World Congress on the Cornea III, New York, Raven Press, 1988:395-398
- [Background] Stark WJ, Stulting RD, Meyer RF, Foulks GN, Smith RE, Chandler JW, Maguire MG, Bias WB. Sharing tissue typing information from the collaborative corneal transplantation studies. Arch Ophthalmol. 1989 May;107(5):633. doi: 10.1001/archopht.1989.01070010651004. No abstract available. PMID 2655566
- [Background] The collaborative corneal transplantation studies (CCTS). Effectiveness of histocompatibility matching in high-risk corneal transplantation. The Collaborative Corneal Transplantation Studies Research Group. Arch Ophthalmol. 1992 Oct;110(10):1392-403. PMID 1417537
- [Background] McDonnell PJ, Enger C, Stark WJ, Stulting RD. Corneal thickness changes after high-risk penetrating keratoplasty. Collaborative Corneal Transplantation Study Group. Arch Ophthalmol. 1993 Oct;111(10):1374-81. doi: 10.1001/archopht.1993.01090100082032. PMID 8216018
- [Background] Fink N, Stark WJ, Maguire MG, Stulting D, Meyer R, Foulks G, Smith RE, Rapoza P. Effectiveness of histocompatibility matching in high-risk corneal transplantation: a summary of results from the Collaborative Corneal Transplantation Studies. Cesk Oftalmol. 1994 Feb;50(1):3-12. PMID 8137435
- [Background] Maguire MG, Stark WJ, Gottsch JD, Stulting RD, Sugar A, Fink NE, Schwartz A. Risk factors for corneal graft failure and rejection in the collaborative corneal transplantation studies. Collaborative Corneal Transplantation Studies Research Group. Ophthalmology. 1994 Sep;101(9):1536-47. doi: 10.1016/s0161-6420(94)31138-9. PMID 8090456
- [Background] Hahn AB, Foulks GN, Enger C, Fink N, Stark WJ, Hopkins KA, Sanfilippo F. The association of lymphocytotoxic antibodies with corneal allograft rejection in high risk patients. The Collaborative Corneal Transplantation Studies Research Group. Transplantation. 1995 Jan 15;59(1):21-7. doi: 10.1097/00007890-199501150-00005. PMID 7839424
- [Background] Kamp MT, Fink NE, Enger C, Maguire MG, Stark WJ, Stulting RD. Patient-reported symptoms associated with graft reactions in high-risk patients in the collaborative corneal transplantation studies. Collaborative Corneal Transplantation Studies Research Group. Cornea. 1995 Jan;14(1):43-8. PMID 7712736